CLINICAL TRIAL: NCT04695574
Title: Development, Reliability and Validity of the Closed Kinetic Chain Lower Extremity Stability Test (CKCLEST): A New Clinical Performance Test
Brief Title: The Closed Kinetic Chain Lower Extremity Stability Test (CKCLEST): A New Clinical Performance Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Halime ARIKAN, Research Assistant, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-029
Record Dates: First submitted 2021-01-01; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Endurance; Lower limb; Performance test; Power; Reliability and Validity; Strength

STUDY DESIGN:
Intervention Model Description: Three-blinded, cross-sectional, repeated-measures clinical measurement reliability trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteer young adults (Experimental): Healthy young adults
  Interventions: Procedure: Some clinical evaluation performance tests together with procedure of Closed Kinetic Chain Lower Extremity Stability Test

INTERVENTIONS:
Procedure: Some clinical evaluation performance tests together with procedure of Closed Kinetic Chain Lower Extremity Stability Test — Clinical evaluation methods
  Other Names: Vertical Jump Test; Isokinetic Dynamometer Test; Single Leg Hop Test; Prone Bridge Test

SUMMARY:
It becomes important to evaluate closed kinetic chain activity. The aim of this study was to develop and to determine the test-retest, intra- and interreliability, and validity of the Closed Kinetic Chain Lower Extremity Stability Test (CKCLEST).

DETAILED DESCRIPTION:
Closed kinetic chain activities and exercises are used more and more in rehabilitation programs as they take place in daily life as functional movements. Therefore, it becomes important to evaluate closed kinetic chain activity. The aim of this study is to develop and to determine the test-retest, intra- and interreliability, and validity of the Closed Kinetic Chain Lower Extremity Stability Test (CKCLEST). Three-blinded, cross-sectional, repeated-measures clinical measurement reliability trial. To assess the reliability of CKCLEST, intraclass correlation coefficient (ICC), standard error of measurement (SEM), minimal detectable change (MDC), and Bland-Altman plot will be used. For concurrent validity of CKCLEST will be applied Spearman correlation analysis with Vertical Jump Test, Isokinetic Dynamometer Test, Single Leg Hop Test, and Prone Bridge Test. All analyses were made for both the best score and the average score. This test allows the evaluation of functional lower extremity stability, static/dynamic control of the lower extremity (knee/hip) or trunk, and simultaneous activation of the quadriceps and hamstring muscles / such coactivation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who healthy adults,
* Volunteer

Exclusion Criteria:

* Surgery last six months and pain,
* Disability,
* Instability,
* Limited range of motion in knee function,
* Chronic diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
To determine the concurrent validity of the Closed Kinetic Chain Lower Extremity Stability Test (CKCLEST) | 45 minutes
  For concurrent validity of CKCLEST was applied Spearman correlation analysis with Vertical Jump Test, Isokinetic Dynamometer Test, Single Leg Hop Test, and Prone Bridge Test.

SECONDARY OUTCOMES:
To determine the the test-retest, intra- and interrater reliability of the Closed Kinetic Chain Lower Extremity Stability Test (CKCLEST) | 4 minutes, 7-14 days apart.
  To assess the reliability of CKCLEST, it was applied twice.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University, Ankara
  - Halime ARIKAN, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: No
The study does not contain any patient records and numbers. Individuals are healthy and they filled out the informed consent form.